CLINICAL TRIAL: NCT04860804
Title: A Comparison of Proprietary Formulations of Oral Ketamine + Aspirin and Oral Ketamine Alone in Adult Patients Presenting to the ED With Acute Musculoskeletal Pain: Prospective, Randomized, Open-Label, Clinical Trial.
Brief Title: A Comparison of Proprietary Formulations of Oral Ketamine + Aspirin and Oral Ketamine Alone for Musculoskeletal Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02-02-MMC
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Pain
Keywords: Emergency Medicine, Pain, Pain Management, Musculoskeletal; Emergency Medicine; Pain; Pain Management; Musculoskeletal
MeSH Terms: conditions — Pain; Agnosia | interventions — Aspirin; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AOK Group (Active Comparator): Drug: Proprietary oral formulation of 0.5mg/kg of ketamine + 324mg of aspirin
  Interventions: Drug: Aspirin and Ketamine
- OK Group (Active Comparator): Drug: Proprietary oral formulation of 0.5mg/kg of ketamine
  Interventions: Drug: Oral Ketamine

INTERVENTIONS:
Drug: Aspirin and Ketamine — Drug: Proprietary oral formulation of 0.5mg/kg of ketamine + 324mg of aspirin
  Arms: AOK Group
Drug: Oral Ketamine — Proprietary oral formulation of 0.5mg/kg of ketamine
  Arms: OK Group

SUMMARY:
Acute Pain is one of the most frequent chief complaints and the main reason for visiting the Emergency Department (ED). The acute pain in the ED is largely prevalent across the country with recent literature demonstrating that 61-91% of patients are admitted to the ED due to a variety of acute painful syndromes. There is a lack of good options for pain control in such settings.

DETAILED DESCRIPTION:
STUDY OBJECTIVES: To compare analgesic efficacy and rates of side effects of a proprietary formulation of orally administered aspirin and ketamine (AOK) to a proprietary formulation of Oral Ketamine (OK) (VTS-K formulations) for pain management in adult ED patients presenting to the ED with acute musculoskeletal pain HYPOTHESIS: The investigators hypothesize that the administration of AOK will provide better analgesia at 60 minutes post-administration in comparison to OK in adult patients presenting to the ED with acute musculoskeletal pain. The primary outcome of this trial is the comparative reduction in participant's pain scores at 60 minutes post-medication administration.

STUDY DESIGN:

Subjects: Patients 18 years of age and older presenting to the ED with acute musculoskeletal painful conditions (traumatic and non-traumatic) with an initial pain score of 5 or more on a standard 11-point (0 to 10) numeric rating scale and requiring oral analgesia as determined by the treating attending physician. Patients' screening and enrollment will be performed by study investigators and research assistants. All patients will be enrolled at various times of the day when study investigators will be available for patient enrollment and an ED pharmacist will be available for medication preparation.

Design: This is a prospective, randomized, open-label trial comparing analgesic efficacy and safety of AOK and OK in patients presenting to the ED of Maimonides Medical Center with acute musculoskeletal pain. Upon meeting the eligibility criteria, patients will be randomized into one of the two study arms: Group I will receive AOK and Group II will receive OK.

Data Collection Procedures: Each patient will be approached by a study investigator for acquisition of written informed consent and Health Insurance Portability and Accountability Act authorization after being evaluated by the treating emergency physician and determined to meet study eligibility criteria. When English will not be the participant's primary language, a language- appropriate consent form will be used and non-investigator, hospital employed, trained interpreters or licensed telephone interpreters will assist in acquisition of informed consent. Baseline pain score will be determined with an 11-point numeric rating scale (0 to 10), described to the patient as "no pain" being 0 and "the worst pain imaginable" being 10. A study investigator will record the patient's body weight and baseline vital signs. All data will be recorded on data collection sheets, including patients' sex, demographics, medical history, and vital signs, and entered into SPSS (version 24.0; IBM Corp) by the research manager. Confirmation of written consent acquisition for all participants, and statistical analyses will be conducted by the statistician, who will work independently of any data collection.

Expected Outcomes: The primary outcome will include a reduction from baseline of pain scores on numeric rating pain scale (NRS) at 60 minutes. The secondary outcomes will include a need for rescue analgesia and rates of adverse up to 120 minutes. With respect to unique adverse effects of SDK, we will use Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) and Richmond Agitation Sedation Scale (RASS). SERSDA Scale includes fatigue, dizziness, nausea, headache, feeling of unreality, changes in hearing, mood change, general discomfort, and hallucinations with severity of each graded by patients on a five-point scale, with "0" representing the absence of any adverse effects and "4" representing a severely bothersome side effect. RASS evaluates the severity of agitation and/or sedation in accordance to the nine-point scale with scores ranging from "-4" (deeply sedated) to "0" (alert and calm) to "+4" (combative).

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older
* acute musculoskeletal pain
* initial pain score of 5 or more on a standard 11- point (0 to 10) numeric rating scale.
* awake, alert, and oriented to person, place, and time

Exclusion Criteria:

* altered mental status,
* allergy to aspirin and ketamine,
* pregnant
* unstable vital signs (systolic blood pressure <90 or>180 mm Hg, pulse rate <50 or >150 beats/ min, and respiration rate <10 or >30 breaths/min)
* inability to provide consent
* consumption of Aspirin or NSAID's within 6 hours of arrival to the ED
* active PUD
* history of GI Hemorrhage
* history of renal and hepatic insufficiency
* past medical history of alcohol or drug abuse
* schizophrenia

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leily Naraghi Bagher Pour, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerges L, Fassassi C, Barberan C, Correa Bravo S, Davis A, Drapkin J, Likourezos A, Silver M, Hossain R, Niceforo P, Gohel A, Motov S. Oral Aspirin/ketamine versus oral ketamine for emergency department patients with acute musculoskeletal pain. Am J Emerg Med. 2022 Aug;58:298-304. doi: 10.1016/j.ajem.2022.05.026. Epub 2022 May 19. PMID 35777275

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AOK Group | OK Group
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AOK Group | OK Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 16 | 20 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score at 60 Minutes
Description: Change of pain scores on numeric rating pain scale (NRS) at 60 minutes mark form the baseline. The NRS is an 11 item Likert Scale ranging from 0 (no pain) to 10 (very severe pain) with 5 indicating moderate pain.
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AOK Group | OK Group
Number analyzed (Participants) | 28 | 28
units on a scale | 2.18 (2.1) | 4.01 (2.1)

ADVERSE EVENTS:
Time Frame: 60 minutes
Arm/Group | AOK Group | OK Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT04860804/Prot_SAP_000.pdf